CLINICAL TRIAL: NCT01939483
Title: A Pilot Study of Irinotecan in Patients With Breast Cancer and CNS Metastases
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Rita Sanghvi, Mehta, HS Clinical Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 11-22; 2011-8497 (Other: University of California, Irvine); NCI-2013-01136 (Other: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2013-09-06; First posted 2013-09-11 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Central Nervous System Metastases; Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
Keywords: Irinotecan hydrochloride; Irinotecan; CAMPTOSAR
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (irinotecan hydrochloride) (Experimental): Patients receive irinotecan hydrochloride IV over 90 minutes on days 1, 8, 15, 22, and 29. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  This arm also includes laboratory biomarker analysis as an intervention.
  Interventions: Drug: irinotecan hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; camptothecin-11; CPT-11; irinotecan; irinotecan HCl; U-101440E
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies irinotecan hydrochloride in treating patients with breast cancer and brain metastases that progressed after whole brain radiation therapy or stereotactic radiosurgery. Drugs used in chemotherapy, such as irinotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES; I. To evaluate the safety and efficacy of irinotecan (irinotecan hydrochloride) in breast cancer patients with brain metastases who progressed after radiation therapy.

II. To estimate central nervous system (CNS) objective response and clinical benefit rate in patients with breast cancer and brain metastases treated with irinotecan.

III. To estimate progression free survival. IV. To estimate overall survival. V. To assess the toxicity of Irinotecan.

OUTLINE:

Patients receive irinotecan hydrochloride intravenously (IV) over 90 minutes on days 1, 8, 15, 22, and 29. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of breast cancer (irrespective of receptor status), with evidence of CNS disease by computed tomography (CT) or magnetic resonance imaging (MRI), who have progressed after whole brain radiation therapy or stereotactic radiosurgery
* Patients must not be a candidate for surgical resection and/or further stereotactic radiosurgery
* Patients may have had an unlimited number of prior treatments, including any systemic chemotherapy (excluding prior progression of disease with topoisomerase inhibitors as explained below), surgical resection, whole brain radiation, stereotactic radiosurgery, or radioimmunotherapy
* Patient must have MRI of brain obtained within two weeks of study initiation for staging and patients must also receive first dose within two weeks of study enrollment
* Patients must have at least one measurable brain lesion prior to start of treatment (≥ 10 mm on T1-weighted, gadolinium-enhanced MRI)
* Karnofsky performance score greater than 60
* At least two weeks must have elapsed since prior chemotherapy, three weeks must have elapsed since last surgery, and six weeks since completion of radiation therapy
* Hemoglobin > 9
* Absolute neutrophil count (ANC) > 1500
* Platelet count (plt) > 125
* Creatinine < 1.5
* Total bilirubin < 1.5
* Aspartate aminotransferase and alanine aminotransferase levels within five times the upper limit of normal
* Patients may be on oral corticosteroids at stable dose (no dose change within two weeks of enrollment), and may be on antiepileptic medication (except for cytochrome P450 3A4 (CYP3A4) enzyme-inducing antiepileptic medications)
* Fertile patients must use effective contraception

Exclusion Criteria:

* Pregnancy, lactation, immunosuppression other than corticosteroids
* Patient may be on hormonal therapy or Herceptin, but no other concurrent chemotherapy is allowed
* Patients who had progression of their breast cancer after prior administration of irinotecan are excluded
* Patients with leptomeningeal carcinomatosis as the only site of CNS involvement are excluded
* No other active malignancy except for any of the following: curatively treated basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, other malignancies considered disease-free
* Patients using valproic acid within the last two weeks and patients with contraindications to anticholinergic agents will be excluded
* Concurrent administration of CYP3A4 enzyme-inducing antiepileptic medications (e.g. phenytoin) will not be allowed (if patients are taking one of these agents, they must switch to a non- enzyme-inducing antiepileptic medication prior to start of treatment)
* No history of immediate or delayed-type hypersensitivity reaction to gadolinium contrast agents or other contraindication to gadolinium contrast, and no other known contraindication to MRI
* Homozygous for uridine diphosphate (UDP) glucuronosyltransferase 1 family, polypeptide A1 (UGT1A1)*28 allele * All patients will be tested for UGT1A genotype prior to starting treatment and be excluded if they are homozygous for the UGT1A1*28 allele (UGT1A1 7/7 genotype); irinotecan's active metabolite glucuronidation of 7-ethyl-10-hydroxycamptothecin (SN-38) is inactivated through glucuronidation by uridine diphosphate glucuronosyltransferases (UGTs) mainly in the liver and is excreted through the bile ducts; a meta-analysis demonstrated that the UGT1A1*28 genotype is moderately predictive of severe irinotecan induced hematologic toxicity at moderate doses and strongly predictive at high doses, and in 2005, the Food and Drug Administration (FDA) added a warning to the irinotecan packaging label that patients with the UGT1A1*28 genotype were at increased risk for neutropenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2017-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
CNS objective response (complete response or partial response), defined as at least 20% volumetric reduction of CNS lesions in absence of increasing steroid use, progressive neurologic signs and symptoms, or progressive extra-CNS disease, based on MRI | Up to 24 months
Response rate of patients who have remained progression-free, based on MRI | Up to 6 months

SECONDARY OUTCOMES:
Overall survival | Time between treatment initiation and death, assessed up to 24 months
  The product limit estimator developed by Kaplan and Meier was used to graphically describe the distribution of survival among patients with recurrent disease.
Progression free survival (PFS) | Time between treatment initiation and disease progression/relapse/death, assessed up to 24 months
  The product limit estimator developed by Kaplan and Meier was used to graphically describe the distribution of PFS among patients with recurrent disease.
Clinical benefit rate (objective response + stable disease at least 16 weeks) | Up to 24 months
Frequency of toxicity occurrence, assessed by National Cancer Institute's Common Terminology Criteria (CTC) for Adverse Events version 4.0 | Up to 24 months
  Tabulated by type, and worst grade experienced by the patient. Toxicity will initially be summarized within each cohort or patient subgroup, and then collectively summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Mehta, MD, Principal Investigator — University of California, Irvine